CLINICAL TRIAL: NCT05010876
Title: Evaluation of the Effects of Bradykinin Antagonists on Pulmonary Manifestations of COVID-19 Infections (AntagoBrad-Cov Study).
Acronym: AntagoBrad
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-002225-29
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Complement C1 Inhibitor Protein; icatibant

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, multicentre, prospective study of three parallel groups of patients.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- standard care + C1 inhibitor (Experimental): The C1 inhibitor will be used at a dose of 1000 units per slow infusion (two hours). Two infusions will be given 24 hours apart. These doses correspond to the usual doses used in the treatment of conditions in which the C1-Inhibitor is indicated.
  Interventions: Drug: C1 Inhibitor Human; Other: Placebo
- standard care + Icatibant + C1 inhibitor (Experimental): The C1 inhibitor will be used at a dose of 1000 units per slow infusion (two hours). Two infusions will be given 24 hours apart. These doses correspond to the usual doses used in the treatment of conditions in which the C1-Inhibitor is indicated.
  The icatibant will be used in a single injection of 30 mg subcutaneously, preferably in the abdominal region. These doses correspond to the doses usually used in the treatment of conditions in which icatibant is indicated.
  Interventions: Drug: C1 Inhibitor Human; Drug: Icatibant Injection
- standard care + placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: C1 Inhibitor Human — standard care + 1000 units of C1 inhibitor during 2 slow infusions of 500 units
  Arms: standard care + C1 inhibitor; standard care + Icatibant + C1 inhibitor
Drug: Icatibant Injection — a single injection of 30 mg subcutaneously
  Arms: standard care + Icatibant + C1 inhibitor
Other: Placebo — The placebo will be physiological serum presented in forms mimicking the C1-Inhibitor and the icatibant.
  Arms: standard care + C1 inhibitor; standard care + placebo

SUMMARY:
The main objective of this study is to evaluate the efficacy of human C1 inhibitor, administered alone or in combination with icatibant (a specific bradykinin B2 receptor antagonist) on the pulmonary manifestations of COVID-19 infections.

DETAILED DESCRIPTION:
Prospective, prospective, multicentre, double-blind, randomised, multi-centre study of three parallel groups of patients:

* Group 1 (n=15): standard of care + C1 inhibitor
* Group 2 (n=15): standard care + icatibant + C1 inhibitor
* Group 3 (n=15): standard support + placebo

The study has two parts:

* A 4-day (96-hour) therapeutic part during which the patient will be evaluated nine times (H0, H4, H12, H24, H36, H48, H60, H72 and H96).
* A follow-up part of 6 days with at least two assessments (D7 and D10).

The maximum duration of patient participation in the study will be 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age, having read and signed the consent form for participation in the study after the reflection period (≤ 15 minutes)
* Patient screened for COVID+ by RT-PCR on nasopharyngeal swab
* Patient with at least three of the following respiratory signs:

  * Temperature >38° C
  * Non-productive dry cough
  * Presence of crackling rales on auscultation
  * Respiratory discomfort felt by the patient
  * Heart rate > 90/min
  * Respiratory rate >20/min
  * O2 saturation ≤ 93%
* Patient whose clinical condition, in the opinion of the investigator, requires hospital monitoring.
* Patient who would have been monitored and treated outside of study participation, including prevention of thromboembolic risk with LMWH.

Exclusion Criteria:

* Patient with pre-existing respiratory disease (cancer, COPD, asthma, emphysema) or smoking history of > 25 years)
* Patient with a known allergy to one of the study products
* Patient treated with anti TNF, IL1 or IL6
* Patient requiring immediate intubation
* Patient on a low sodium diet
* Patient under protective custody, guardianship or trusteeship
* Patient not affiliated to the French social security system
* Patient participating in another therapeutic protocol
* Pregnant or likely to become pregnant (woman of childbearing age without effective contraception and without HCG dosage)
* Patient unable to understand informed information and/or give written informed consent: dementia, psychosis, consciousness disorders, non-French speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation respiratory discomfort | 96 hours after the administration of treatment
  To evaluate the efficacy of human C1 inhibitor, administered alone or in combination with icatibant (a specific bradykinin B2 receptor antagonist) on the pulmonary manifestations of COVID-19 infections.
  The evaluation of the treatment efficacy of the study is based on the clinical monitoring of the patient and particularly on the following combination of criteria as experienced by the patient :
  * no respiratory discomfort
  * heart rate between 60 and 90 /min
  * respiratory rate less than 20/min
  * O2 saturation greater than 94% without oxygen supply
Efficacy evaluation heart rate between 60 and 90 /min | 96 hours after the administration of treatment
  To evaluate the efficacy of human C1 inhibitor, administered alone or in combination with icatibant (a specific bradykinin B2 receptor antagonist) on the pulmonary manifestations of COVID-19 infections.
  The evaluation of the treatment efficacy of the study is based on the clinical monitoring of the patient and particularly on the following combination of criteria as experienced by the patient :
  * no respiratory discomfort
  * heart rate between 60 and 90 /min
  * respiratory rate less than 20/min
  * O2 saturation greater than 94% without oxygen supply
Efficacy evaluation respiratory rate less than 20/min | 96 hours after the administration of treatment
  To evaluate the efficacy of human C1 inhibitor, administered alone or in combination with icatibant (a specific bradykinin B2 receptor antagonist) on the pulmonary manifestations of COVID-19 infections.
  The evaluation of the treatment efficacy of the study is based on the clinical monitoring of the patient and particularly on the following combination of criteria as experienced by the patient :
  * no respiratory discomfort
  * heart rate between 60 and 90 /min
  * respiratory rate less than 20/min
  * O2 saturation greater than 94% without oxygen supply
Efficacy evaluation O2 saturation greater than 94% without oxygen supply | 96 hours after the administration of treatment
  To evaluate the efficacy of human C1 inhibitor, administered alone or in combination with icatibant (a specific bradykinin B2 receptor antagonist) on the pulmonary manifestations of COVID-19 infections.
  The evaluation of the treatment efficacy of the study is based on the clinical monitoring of the patient and particularly on the following combination of criteria as experienced by the patient :
  * no respiratory discomfort
  * heart rate between 60 and 90 /min
  * respiratory rate less than 20/min
  * O2 saturation greater than 94% without oxygen supply

SECONDARY OUTCOMES:
Tolerance evaluation | Day 10
  The tolerance of the study products will be assessed by collecting adverse events that occurred during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Denis VINCENT, MD PD, Study Director — Médecine interne, Faculté de Montpellier
Locations (1):
- Hôpital Privé de Parly II, Le Chesnay, France